CLINICAL TRIAL: NCT06762067
Title: Exercise Training in Front of a Mirror for Intermittent Exotropia Control Post Strabismus Surgery: A Randomized Controlled Study
Brief Title: Exercise Training on a Mirror for Intermittent Exotropia Control Post Strabismus Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Nawwar Abdallah KHattab, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nesma-005418
Record Dates: First submitted 2024-12-23; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Exercise Training; Intermittent Exotropia; Strabismus
MeSH Terms: conditions — Strabismus | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirror therapy (Experimental): It will include 20 patients. They will receive traditional physical therapy exercise using mirror therapy twice a week ,for 3 months ,and subjects will do the same exercise at home daily with the aid of mother and level of adherence will be checked every session
  Interventions: Other: mirror therapy
- Traditional therapy (Active Comparator): It will include 20 patients. They will receive traditional physical therapy exercise only twice a week ,for 3 months ,and subjects will do the same exercise at home daily with the aid of mother and level of adherence will be checked every session
  Interventions: Other: traditional therapy

INTERVENTIONS:
Other: mirror therapy — Participants will undergo physiotherapy exercises in a mirror alongside post-surgery care. The program includes palming exercises, eye exercises, pencil push-ups, Brock string exercises, thumb exercises, and proprioceptive neuromuscular facilitation exercises. The first exercise warms up extra ocular muscles, the second improves eye coordination, the third motivates the lazy eye, the fourth strengthens eye muscles, and the fifth involves a near-distance jump for oblique muscles.
  Arms: Mirror therapy
Other: traditional therapy — The patients within the control group will receive traditional care post-strabismus operation as eye glasses and eye drops and regular exercise
  Arms: Traditional therapy

SUMMARY:
The study aims to explore the impact of mirror therapy on exodeviation control, near and far strabismus angles, and quality of life in intermittent exotropia control post strabismus surgery, as well as its effects on near and far strabismus angles.

DETAILED DESCRIPTION:
Strabismus is a common childhood disorder causing eye deviation, affecting life quality and cosmetic appearance. Early detection and management improve binocular function and psychosocial problems. Intermittent exotropia is a common type. Surgery is the most common method for correcting strabismus, but complications can be difficult to treat. Physical therapy programs are limited in treating strabismus after surgery, and adding mirror therapy to traditional treatments may help maintain surgery results. This thesis aims to decrease this knowledge gap and improve the treatment of strabismus.

ELIGIBILITY:
Inclusion Criteria:

1. 40 boys and girls with ages from 5 to 15 years
2. History of strabismus surgery from 6 months presence of intermittent exotropia.
3. Normal sensory and motor fusion, equal visual acuity. Good general health condition.
4. Ability to understand and do the exercises at home

Exclusion Criteria:

1. systemic diseases as myasthenia gravis, multiple sclerosis and diabetes
2. Optic nerve injury, organic ocular disease, attention disorder and mental disorders
3. Attention disorder and learning disability

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of change of the exodeviation control | at baseline and after 3 months
  The ophthalmologist examines participants' eyes while focusing on an accommodative target, determining their exotropia score. The scores range from constant to dissociated, with no exotropia unless dissociated and maximum score is 5 and minimal score is 0. the lower score is the better

SECONDARY OUTCOMES:
Assessment of change of the near strabismus angles | at baseline and after 3 months
  the near strabismus angles will be measured by using prisms of different powers
Assessment of change of the far strabismus angles | at baseline and after 3 months
  The prism cover test is a method used to measure the angle of deviation of a small-angle tropia. It involves covering the non-fixating eye with a prism oriented in the same direction as the deviation, blocking the fixating eye simultaneously. The strength of the prism is adjusted to prevent fixation shift and reduce deviation. Near and far strabismus angles are measured using prisms of varying powers. The measurement should be taken at 33 cm, 6 m, and occasionally at 60 m, and with or without corrective lenses.
Assessment of change of questions of Child and Proxy health related quality of life | at baseline and after 3 months
  The final Child and Proxy health-related quality of life questionnaires for intermittent exotropia are designed to gather information about the concerns and difficulties faced by children and adolescents with this condition. The questionnaires are formatted for 5-7-year-old children, 8-17-year-old children, and PROXY children.
Assessment of change of questions of health-related quality of life questionnaire for Parents of children with intermittent exotropia | at baseline and after 3 months
  Parents of children with intermittent exotropia often express concerns about their child's eyesight, including potential physical and psychological effects.